CLINICAL TRIAL: NCT01112761
Title: Cortical Plasticity Assessment in Athletes With a History of Concussion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources to run the trial
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010P000191
Record Dates: First submitted 2010-04-20; First posted 2010-04-28 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Concussion
Keywords: Athletes; Multiple Concussions; Transcranial Stimulation
MeSH Terms: conditions — Brain Concussion | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Subjects (Experimental): Each subject will undergo each of the three conditions (active anodal tDCS, cathodal tDCS and sham tDCS), but the order in which they do so will be randomized.
  Interventions: Device: Transcranial direct current stimulation
- Athletes with history of concussion (Experimental): Each subject will undergo each of the three conditions (active anodal tDCS, cathodal tDCS and sham tDCS), but the order in which they do so will be randomized.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Each type of stimulation will be administered with a time interval of a week in between to prevent any carryover affects.

SUMMARY:
The purpose of this research is to determine whether athletes with concussion have changes in cortical excitability.

Single and paired transcranial magnetic stimulation (TMS) can be used as reliable neurophysiological marker of motor cortex reorganization in athletes with concussions.

This study also aims to determine whether modulation of cortical activity by a powerful technique of noninvasive brain stimulation (tDCS) results in a different cortical response as compared with sham tDCS.

DETAILED DESCRIPTION:
This study is a multicenter study with investigators from other institutions (Dr. Alvaro Pascual-Leone and Dr. Hugo Theoret).

ELIGIBILITY:
Inclusion Criteria:

* Student-athletes at risk for traumatic brain injury (collegiate football, ice hockey)
* Age between 18 and 30 yr.
* Concussion as defined by the American Academy of Neurology: trauma-induced alteration in mental status that may or may not involve loss of consciousness (confusion and amnesia are the hallmarks of concussion)
* Concussion that occurred > 6 months
* All head injuries classified as minor with a Glasgow Coma Scale of 13 to 15 at the time of the trauma
* Participants are cleared for full sport participation based upon neurological and neuropsychological (NS) assessments Classified as symptomatic based on Post-concussion Symptom List

Exclusion Criteria:

* Previous significant neurological history
* Use of tricyclic anti-depressants such as amitriptyline, nortriptyline and imipramine within the past six months.
* Use of anticonvulsants such as carbamazepine, phenytoin, valproic acid and gabapentin within the past six months
* History of seizures, depression or PTSD
* Presence of post-concussion symptoms such as complaints of loss of concentration, dizziness, fatigue, headache, irritability, visual disturbances, and light sensitivity.
* Contraindications to single pulse TMS (TMS will be used to measure cortical excitability) such as metal head implants
* history of seizures
* unexplained loss of consciousness
* metal in the head
* frequent or severe headaches or neck pain
* implanted brain medical devices.
* Contraindications to tDCS:
* metal in the head
* implanted brain medical devices

For the control group (subjects with no concussion) we will select subjects according to the previously stated list of exclusions as well as the following criteria: Subjects who are athletes (similar to the concussed group) with the same age range and also similar level of education; however these subjects will have no prior history of concussion or neurological insult as self reported. They should also have no contraindications to TMS or tDCS.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Cortical excitability and cortical plasticity assessment | Baseline, 1st, 2nd and 3rd week
  TMS and tDCS

SECONDARY OUTCOMES:
Cognitive functioning in athletes with concussion compared to athletes without concussion | Baseline, 1st, 2nd and 3rd week
  Will use the Immediate Postconcussion Assessment and Cognitive Test (IMPACT): a neuropsychological test battery that measures aspects of cognitive functioning including attention, memory, reaction time and information processing speed.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States